CLINICAL TRIAL: NCT01752647
Title: Cohort Study of Low Dose Computed Tomography for Lung Cancer Screening in Asymptomatic High-risk Patients.
Brief Title: CT Screening For Lung Cancer in High Risk Patients: the Russian Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RLCT-01
Record Dates: First submitted 2012-12-13; First posted 2012-12-19 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer
Keywords: lung cancer; screening; low dose; computed tomography
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low dose computed tomography (Experimental): Patients will have one baseline LDCT scan.
  Interventions: Procedure: Low dose computed tomography

INTERVENTIONS:
Procedure: Low dose computed tomography — Low dose computed tomography scan
  Other Names: CT scan; LDCT scan

SUMMARY:
This prospective cohort trial was planned to assess the feasibility of establishing a lung cancer screening program in Russian Federation using low-dose CT scanning in asymptomatic patients with at least a 30 pack-year history of cigarette smoking.

DETAILED DESCRIPTION:
Low dose computer tomography (LDCT) showed promising results in recently published studied. Lung cancer screening programs with fluorography introduced in USSR in 70s-80s showed shift to earlier stages with no data on mortality. No other studies or programs on lung cancer screening were introduced in Russia since then.

The purpose of this study is to assess the feasibility of establishing a lung cancer screening program in Russian Federation using LDCT scanning in asymptomatic patients with at least a 30 pack-year history of cigarette smoking. This cohort prospective study is planned to enroll at least 500 current or former smokers.

Patients will be screened by LDCT scan at baseline with recommendation to perform follow-up in case of any positive result. For nodes more than 10 mm full clinical examination is recommended. For nodes 3-9.9 mm follow-up scans in 1, 3 or 6 months is recommended. For nodes smaller than 3 mm and negative results annual LDCT is recommended. Patient with positive results will be followed until final clinical diagnosis.

Secondary outcomes include:

* Lung cancer diagnoses
* Lung cancer and overall mortality
* Quality of life assessment
* Complications of diagnostic and surgical procedures following a positive result.
* Comparison of independent radiological evaluation of scans.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years
* 30 or more pack-years of cigarette smoking history
* Former smokers: quit smoking within the previous 10 years
* Ability to tolerate CT procedure
* Signed informed consent

Exclusion Criteria:

* Any cancer other than nonmelanoma skin cancer or carcinoma in situ in the 5 years prior to eligibility assessment
* Severe uncontrolled heart, vascular, respiratory or endocrine pathology.
* Life-expectancy less than 1 year
* History of lung cancer
* History of lung surgery.
* Acute respiratory disease
* Hemoptysis.
* Weight loss more than 10 kg in the 12 months prior to eligibility assessment
* Participation in other cancer clinical trial
* Chest CT examination in the 12 months prior to eligibility assessment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Estimate the time period for recruitment of 500 participants in LDCT screening study. | 3 months
  Primary outcome measure is to assess the feasibility of establishing a lung cancer screening program in Russian Federation using low-dose CT scanning in asymptomatic patients with at least a 30 pack-year history of cigarette smoking. The main concern comes from the possibility to recruit participant for screening as small amount of information is available about lung cancer screening options for high-risk population and general practitioners in different regions of the country.

SECONDARY OUTCOMES:
Lung cancer detection rate | One year
  Assess number of lung cancer diagnoses after radiological and morphological verification of positive lung nodules.
All-cause mortality | 5 years
  Assess all-cause mortality mortality within next 5 years.
Lung cancer mortality | 5 years
  Assess lung cancer mortality in the screened group within next 5 years.
Nodule detection rate | 3 months
  Estimate nodule detection rate, types and sizes of lung nodules found.
Recruitment strategies | 3 months
  Assess the efficacy of different recruitment strategy in this study. Information about the study was shared between general practitioners, radiologists, pulmonologists, thoracic oncologist.

OTHER OUTCOMES:
Comparison of independent radiological evaluation of scans | One year
  Comparison of independent radiological evaluation of scans performed by 2 independent specialists.
Lung nodules management | 12 months
  Assess algorithms for lung nodules management in regional oncology hospitals in Russian Federation.
Frequency of diagnostic procedures. | 12 months
  Estimate the frequency of diagnostic procedures, types of invasive and non-invasive procedures performed.
Complication of diagnostic procedures | 12 months
  Assess the complication rate after diagnostic procedures performed after screening. Procedures include baseline LDCT.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Barchuk, MD PhD, Study Chair — N.N. Petrov National Medical Research Center of Oncology
Locations (2):
- Russia (2):
  - Semashko City Clinical Hospital #2, Samara, Samara Oblast
  - Samara Regional Oncology Dispansery, Samara, Samara Oblast